CLINICAL TRIAL: NCT02367365
Title: Neovascular Morphology and Persistent Disease Activity Among Patients With Neovascular Age-Related Macular Degeneration
Brief Title: Neovascular Morphology and Persistent Disease Activity Among Patients With NV AMD
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00055232
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2017-11

CONDITIONS: Neovascular Age-Related Macular Degeneration
Keywords: Neovascular Age-Related Macular Degeneration; anti-vascular endothelial growth factor; neovascular lesion morphology; indocyanine green angiography; persistent disease activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treatment Naive NVAMD Patients: Patients with treatment naive NVAMD diagnosed in the last three months
  Interventions: Other: No Intervention
- Newly Reactivated NVAMD Patients: Patients with newly reactivated NVAMD which has been previously quiescent off treatment
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention
  Groups: Treatment Naive NVAMD Patients
Other: No Intervention — No intervention
  Groups: Newly Reactivated NVAMD Patients

SUMMARY:
Neovascular Age-Related Macular Degeneration (NV AMD) remains the leading cause of vision loss among people over 65. Intravitreal injections with drugs that block VEGF have revolutionized treatment of NV AMD. However, less than 40% of treated patients have clinically significant imporovement in vision. In this study, we will determine the relative frequency of neovascular subtypes in two groups: 1) a representative, treatment-naive NV AMD patient population, and 2) a population of patients who develop recurrent NV AMD activity while off treatment and assess the frequency of persistent disease activity (PDA) according to specific neovascular morphologic subtypes. This information will clarify the scope of the PDA problem and will identify patients with PDA who may benefit from additional therpeutic strategies.

DETAILED DESCRIPTION:
Neovascular Age-Related Macular Degeneration (NV AMD) remains the leading cause of vision loss among people over 65. Intravitreal injections with drugs that block VEGF, a major protein mediator of angiogenesis and vascular leakage, have revolutionized treatment of NV AMD. However, less than 40% of treated patients have clinically significant improvement in vision. Further, in spite of continuous monthly anti-VEGF therapy, up to 40-50% of patients demonstrate sustained persistent disease activity (PDA), defined as (1) unresolved intraretinal, subretinal, or sub-retinal pigment epithelium fluid; (2) progressive lesion enlargement and fibrosis; and/or (3) persistent or new hemorrhage, assessed after either loading dose therapy or after sustained treatment with anti-VEGF. Since affected patients are at increased risk for long-term vision loss, PDA remains a vital clinical unmet need.

We are interested in the relationship between NV lesion morphology and response to therapy. Specifically, we hypothesize that specific NV morphologic subtypes are more frequently associated with PDA, based on preliminary retrospective analyses of indocyanine green (ICG) imaging data from NV AMD patients in our Duke Medical Retina practice. We have observed that eyes with Capillary pattern, seen as a discrete homogenous focus of microvessels, are highly responsive to anti-VEGF therapy and rarely exhibit PDA (<20% of cases). In contrast, eyes with Arteriolar pattern (large-caliber feeding artery, many branching arterioles, and minimal capillary component) and eyes with polypoidal choroidal vasculopathy (variably sized and numbered, discrete saccular dilations of choroidal vasculature), demonstrate PDA in up to 70% of cases. A third subtype, choroidal leak syndrome, visible as choroidal hyperpermeability and leakage, manifest PDA in over 60% of cases. These data suggest that complex NV lesion morphology is the primary cause of PDA, and that anti-VEGF therapy alone is insufficient for these patients. However, the relative frequency of these subtypes and the association of PDA and NV lesion morphology, in a treatment-naive population free of selection bias, are unknown.

In this study, we will determine the relative frequency of NV subtypes in two groups: (i) a representative, treatment-naïve NV AMD patient population, and (ii) a population of patients who develop recurrent NVAMD activity while off treatment and assess the frequency of PDA according to specific NV morphologic subtypes. This information will clarify the scope of the PDA problem, and will identify patients with PDA who may benefit from additional therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of either treatment naive NVAMD or newly reactivated NVAMD which has been previously quiescent off treatment
* Men and women aged 50 years or older
* Able to provide written informed consent

Exclusion Criteria:

* Potential study eye with ongoing (within previous 6 months of diagnosis of NVAMD disease activity) treatment for CNV, including anti-VEGF medications, corticosteroids, photodynamic therapy, thermal laser photocoagulation, transpupillary thermotherapy, or pneumatic displacement of macular hemorrhage
* CNV secondary to causes other than AMD
* Known or suspected sensitivity or allergy to ICG dye
* Known or suspected sensitivity or allergy to fluorescein dye
* Significant medial opacity (e.g. cataract) precluding clincial imaging adequate for interpretation
* Prior history of vitrectomy surger in potential study eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with treatment naive NVAMD or newly reactivated NVAMD
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2014-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Frequency of ICG neovascular subtypes | 4-6 weeks post loading dose
Percentage of each neovascular subtype exhibiting persistent disease activity | 4-6 weeks post loading dose

CONTACTS AND LOCATIONS:
Overall Officials: Scott Cousins, MD, Principal Investigator — Duke University
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States